CLINICAL TRIAL: NCT00432341
Title: Efficacy and Safety of Two Different Botulinum Toxin Type A Treatments for Moderate to Severe Cervical Dystonia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated early due to difficulties with patient recruitment
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MedAff-BTX-0615
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Results first posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-11

CONDITIONS: Spasmodic Torticollis
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- BOTOX® (Experimental): Botulinum toxin type A (BOTOX®)
  Interventions: Biological: botulinum toxin type A
- Dysport® (Active Comparator): Botulinum toxin type A (Dysport®)
  Interventions: Biological: botulinum toxin type A

INTERVENTIONS:
Biological: botulinum toxin type A — 200 Units at Visit 1 (Day 1)
  Other Names: BOTOX®
  Arms: BOTOX®
Biological: botulinum toxin type A — 500 Units at Visit 1 (Day 1)
  Other Names: Dysport®
  Arms: Dysport®

SUMMARY:
The purpose of this study is to compare two types of botulinum toxin type A to treat the involuntary muscle contractions in the neck

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervical dystonia/spasmodic torticollis for at least 18 months
* Successfully treated previously with botulinum toxin type A

Exclusion Criteria:

* Breast feeding, pregnant, or could become pregnant
* Surgery or spinal cord stimulation for cervical dystonia
* Previous injections of phenol, alcohol for cervical dystonia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- Buenos Aires, Argentina
- Parkville, Victoria, Australia
- New Delhi, New Delhi, India

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOTOX® | Dysport®
Started | 24 | 30
Completed | 24 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BOTOX® | Dysport® | Total
Number analyzed (Participants) | 24 | 30 | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 42.0 (13.1) | 49.9 (12.6) | 46.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Duration of Treatment Benefit
Description: Duration of treatment benefit was measured as the time (days) from Baseline until patients had a loss of therapeutic benefit, as defined by the achievement of their Toronto Western Spasmodic Torticollis Rating Scale Duration Target Score (TDTS) [loss of 80% of benefit].
Time Frame: 20 Weeks
Population: Modified Intent to Treat: included all patients who were randomized to treatment, received treatment at Visit 1, and provided at least 1 post-dose assessment measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 24 | 30
Days | 112.5 [102.0 to 126.0] | 107.0 [102.0 to 118.0]

2. Secondary Outcome: Toronto Western Spasmodic Torticollis Rating Scale Duration Target Score (TDTS) at Week 4
Description: The TDTS was the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) score representing a loss of 80% of the treatment benefit at Week 4. The TDTS is calculated from the TWSTRS score and ranges from 0 (least symptoms) to 68 (worst symptoms). The TWSTRS total score which is scored from 0 (least symptoms) to 85 (worst symptoms).
Time Frame: Week 4
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a Scale
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 24 | 30
Scores on a Scale | 37.0 [16 to 56] | 41.0 [26 to 69]

3. Secondary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Total Score at Week 4
Description: The TWSTRS is an assessment scale used to measure the impact of cervical dystonia on patients. The score is comprised of 3 subscales: Severity, Disability, and Pain, each of which is scored independently. The total of these 3 comprises the TWSTRS total score which is scored from 0 (least symptoms) to 85 (worst symptoms). Higher scores indicate a greater degree of symptom severity.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a Scale
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 24 | 30
Scores on a Scale
  Baseline | 42.0 [17 to 63] | 43.5 [30 to 73]
  Week 4 | 26.0 [10 to 47] | 27.0 [11 to 52]

4. Secondary Outcome: Global Assessment of Benefit by Patient at Week 4
Description: Patient evaluation of benefit from botulinum toxin type A treatment for cervical dystonia. Ratings were on a scale of +4 to -4, with higher scores denoting improvement in cervical dystonia: +4 was 'Complete abolishment of signs and symptoms (about 100% improvement)', 0 represented 'Unchanged', and -4 represented 'Very marked worsening (about 100% worse or greater)'.
Time Frame: Week 4
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 24 | 30
Units on a Scale | 2.0 [0 to 4] | 2.0 [-3 to 3]

5. Secondary Outcome: Global Assessment of Benefit by Physician at Week 4
Description: Physician evaluation of benefit from botulinum toxin type A treatment for cervical dystonia. Ratings were on a scale of +4 to -4, with higher scores denoting improvement in cervical dystonia: +4 was 'Complete abolishment of signs and symptoms (about 100% improvement)', 0 represented 'Unchanged', and -4 represented 'Very marked worsening (about 100% worse or greater)'.
Time Frame: Week 4
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 24 | 30
Units on a Scale | 2.0 [1 to 4] | 2.0 [1 to 3]

6. Secondary Outcome: Physician Assessment of Cervical Dystonia Severity at Week 4
Description: Physician assessment of cervical dystonia severity. The rating was assessed on a scale of 0 to 10, with higher scores denoting greater severity: 0 represented 'No evidence of dystonia' and 10 represented 'Worst cervical dystonia ever'
Time Frame: Baseline, Week 4
Population: Modified Intent to Treat: included all patients who were randomized to treatment, received treatment at Visit 1, and provided as least 1 post-dose assessment measure.
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 24 | 30
Units on a Scale
  Baseline | 7.0 [4 to 9] | 8.0 [4 to 9]
  Week 4 | 4.0 [2 to 6] | 4.0 [1 to 7]

7. Secondary Outcome: Physician Comparison of Benefit to Previous Injections at Week 20
Description: Physicians assessed the improvement in cervical dystonia after the study treatment compared to previous treatment(s) for each patient. Physicians were required to answer "How would you rate the benefit of the current treatment of cervical dystonia with botulinum toxin type A compared to the previous treatment using the following scale?". The response options were 'much worse', 'worse', 'somewhat worse', 'same as previous', 'somewhat better', 'better', and 'much better'.
Time Frame: Week 20
Population: Modified Intent to Treat: included all patients who were randomized to treatment, received treatment at Visit 1, and provided as least 1 post-dose assessment measure. Only completed assessments at this time point are included.
Measure: Number; unit: Number of Responses
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 18 | 24
Number of Responses
  Much Worse | 0 | 0
  Worse | 0 | 1
  Somewhat Worse | 0 | 3
  Same as Previous | 13 | 13
  Somewhat Better | 4 | 5
  Better | 0 | 1
  Much Better | 1 | 1

8. Secondary Outcome: Patient Comparison of Benefit to Previous Injections at Week 20
Description: Patients assessed the improvement in cervical dystonia after receiving the study treatment compared to previous treatment(s). Patients were required to answer "How would you rate the benefit of the current treatment of cervical dystonia with botulinum toxin type A compared to the previous treatment using the following scale?". The response options were 'much worse', 'worse', 'somewhat worse', 'same as previous', 'somewhat better', 'better', and 'much better'.
Time Frame: Week 20
Population: as for outcome 7
Measure: Number; unit: Number of Responses
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 19 | 21
Number of Responses
  Much Worse | 0 | 0
  Worse | 0 | 1
  Somewhat Worse | 0 | 1
  Same as Previous | 8 | 11
  Somewhat Better | 8 | 4
  Better | 0 | 0
  Much Better | 3 | 4

9. Secondary Outcome: Patient Visual Analog Assessment of Pain at Week 4
Description: Patients were required to assess their pain using a Visual Analog Scale in reference to their current perception of pain at that visit. This scale consisted of a line measuring 100 mm, and patients were instructed to put a mark on the line at the point that best described 'How much pain you are having right now'. Higher scores denoted higher pain intensity: 0 indicated 'No pain' and 100 indicated 'Worst possible pain'.
Time Frame: Baseline, Week 4
Population: as for outcome 6
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 24 | 30
Units on a Scale
  Baseline | 49.5 [0 to 81] | 52.0 [0 to 100]
  Week 4 | 20.5 [0 to 58] | 28.0 [0 to 87]

10. Secondary Outcome: Patient Assessment of Need for Retreatment at Week 4
Description: Patients were queried regarding their need for another injection of botulinum toxin type A for cervical dystonia. Patients were required to answer "How would you rate your need for another injection of botulinum toxin type A for cervical dystonia using the following scale?". The response options included 'absolutely requires injection', 'very much requires injection', 'somewhat requires injection', and 'does not require injection'.
Time Frame: Baseline, Week 4
Population: Modified Intent to Treat: included all patients who were randomized to treatment, received treatment at Visit 1, and provided as least 1 post-dose assessment measure. Only completed assessments at the time points are included.
Measure: Number; unit: Number of Responses
Arm/Group | BOTOX® | Dysport®
Number analyzed (Participants) | 23 | 29
Number of Responses
  Absolutely requires injection at Baseline | 19 | 24
  Very much requires injection at Baseline | 5 | 5
  Somewhat requires injection at Baseline | 0 | 0
  Does not require injection at Baseline | 0 | 0
  Absolutely requires injection at Week 4 | 1 | 4
  Very much requires injection at Week 4 | 7 | 5
  Somewhat requires injection at Week 4 | 4 | 3
  Does not require injection at Week 4 | 11 | 17

ADVERSE EVENTS:
Arm/Group | BOTOX® | Dysport®
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/30
Other Adverse Events (participants affected / at risk) | 12/24 | 12/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=24) | Dysport® (N=30)
Dry Mouth (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 1 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulties with patient recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release for a period that is not less than 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication.